CLINICAL TRIAL: NCT01261117
Title: Oral Versus Intravenous Ibuprofen Treatment
Brief Title: Efficacy and Safety of Oral Versus Intravenous Ibuprofen for PDA Treatment in ELBW Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Maternity and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STO5336205575
Record Dates: First submitted 2010-11-29; First posted 2010-12-16 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-11

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent ductus arteriosis; İbuprofen; Extremely Low Birth Weigh infant
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous ibuprofen (Active Comparator): Extremely low birth weight patients receiving iv ibuprofen
  Interventions: Drug: oral ibuprofen
- Oral ibuprofen (Active Comparator): Extremely low birth weight patients receiving oral ibuprofen
  Interventions: Drug: oral ibuprofen

INTERVENTIONS:
Drug: oral ibuprofen — oral or iv ibuprofen in 10, 5 and 5 mg/kg/day with 24 hr intervals

SUMMARY:
To determine whether oral or intravenous ibuprofen has a better or same efficacy and tolerance in closure of patent ductus arteriosis in extremely-low-birth-weight preterm infants.

DETAILED DESCRIPTION:
To determine whether oral or intravenous ibuprofen has a better or same efficacy and tolerance in closure of patent ductus arteriosis in extremely-low-birth-weight preterm infants.Seventy ELBW preterm infants with patent ductus arteriosis will be enrolled in this prospective-randomized study. Patients will receive either intravenous or oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h.

One of the following echocardiographic criteria of a duct size >1.5 mm, a left atrium-to-aorta ratio >1.5, left-to-right shunting of blood, end diastolic reversal of blood flow in the aorta, or poor cardiac function in addition signs of patent ductus arteriosis determined the need of ibuprofen treatment.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight below 1000 gram
* Diagnosed patent ductus arteriosis by Echocardiographic examination

Exclusion Criteria:

* Accompanied other congenital cardiac anomalies
* Severe thrombocytopenia < 60.000
* Severe intracranial bleeding (Grade 3-4)
* Intestinal abnormality and necrotising enterocolitis

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of Oral Versus Intravenous Ibuprofen... ID: STO5336205575 | 6 months
  To compare the closure rate of patent ductus arteriosus after intravenous or oral ibuprofen treatment

SECONDARY OUTCOMES:
Efficacy and Safety of Oral Versus Intravenous Ibuprofen | Results will be identified in 6 months
  Evaluation of renal tolerance and complications

CONTACTS AND LOCATIONS:
Overall Officials: Omer Erdeve, Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)